CLINICAL TRIAL: NCT07255365
Title: VIRTUAL REALITY-BASED 360° CLINIC WALKTHROUGH: EFFECTS ON EXAMINATION ANXIETY AND PHYSICIAN EXAMINATION EASE IN CHILDREN
Brief Title: Virtual Reality-Based 360° Clinic Walkthrough for Reducing Examination Anxiety in Preschool Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Berker Okay (Other)
Responsible Party: Sponsor-Investigator, Berker Okay, MD - Pediatrician (Principal Investigator), Haseki Training and Research Hospital
Organization: Haseki Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 248-2025
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Anxiety; Stress, Psychological; Fear
Keywords: pediatric physical examination; examination anxiety; behavioral distress
MeSH Terms: conditions — Anxiety Disorders; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Children were randomly assigned in a 1:1 ratio to either the virtual reality (VR) pre-examination group or the control group (routine waiting). Both groups underwent the same clinical examination by a blinded pediatrician.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Children and parents were unaware of the study hypothesis. The examining pediatrician and the observer scoring behavioral outcomes were blinded to group allocation. The data analyst also remained blinded until after data lock, ensuring double-blind assessment at evaluator and analyst levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- irtual Reality (VR) Group (Experimental): Children in this arm receive a 3-minute, 360° virtual reality (VR) pre-examination walkthrough of the actual pediatric outpatient clinic using a smartphone-based VR headset. The video presents the waiting area, greeting the pediatrician, and routine non-invasive examination steps from a child's eye-level perspective.
  Intervention(s): Behavioral: Virtual Reality 360° Clinic Walkthrough
  Interventions: Behavioral: irtual Reality 360° Clinic Walkthrough
- Control Group (No Intervention): Children in this arm undergo standard pre-examination waiting without any VR or structured visual preparation. The waiting period is kept similar (approximately 3-5 minutes) to match the duration of the VR exposure.
  Intervention(s): None (routine waiting only)

INTERVENTIONS:
Behavioral: irtual Reality 360° Clinic Walkthrough — A brief, 3-minute 360° video recorded in the actual pediatric outpatient clinic, viewed via VR goggles before examination. The content is child-friendly, non-invasive, and designed to familiarize children with the clinical environment and examination steps to reduce anticipatory anxiety and distress.
  Arms: irtual Reality (VR) Group

SUMMARY:
This prospective, double-blind, randomized controlled trial investigates whether a short, 360° virtual reality (VR) pre-examination walkthrough can reduce anxiety, behavioral distress, and physiological stress responses in preschool children undergoing routine outpatient physical examination. A total of 100 children aged 3-5.5 years were randomized to either a VR group, which viewed a 3-minute real-clinic 360° video via VR goggles, or a control group, which experienced routine waiting only. Primary outcome measures include the Face-Legs-Activity-Cry-Consolability (FLACC) score and crying duration during examination. Secondary outcomes include heart and respiratory rate changes, Wong-Baker Faces Pain Rating Scale (WBS) scores, parent satisfaction, and physician-rated examination ease. The study aims to determine whether immersive, procedure-specific VR preparation can improve examination experience and cooperation while reducing stress for both children and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 5.5 years (36-66 months)
* Clinically stable and presenting for routine outpatient physical examination
* Able to engage with a short audiovisual VR/360° video
* Written informed consent from a parent or legal guardian
* Verbal assent from the child when appropriate

Exclusion Criteria:

* Severe neurodevelopmental delay or communication difficulty
* Autism spectrum disorder or significant behavioral dysregulation
* History of epilepsy or photosensitivity
* Visual or hearing impairment preventing VR use
* Acute illness requiring urgent intervention
* Body temperature ≥ 38.0°C at presentation
* Previous exposure to VR or 360° clinic simulations
* Concomitant sedative medication use
* Refusal of participation by parent or child

Ages: 36 Months to 66 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
FLACC (Face-Legs-Activity-Cry-Consolability) behavioral distress score during examination | During the physical examination (same clinic visit).
  Behavioral distress and pain level during physical examination, assessed using the FLACC scale (score range 0-10; higher scores indicate greater distress).

SECONDARY OUTCOMES:
Crying duration during examination | During the physical examination (same clinic visit).
  Duration of crying (in seconds) recorded with a stopwatch during physical examination; shorter duration reflects lower procedural distress.
Parent satisfaction score | Immediately after the physical examination (same clinic visit).
  Parent-rated satisfaction with the examination process, measured using a 5-point Likert scale (1 = very poor, 5 = excellent).

CONTACTS AND LOCATIONS:
Locations (1):
- SBÜ Sultangazi Haseki Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Escalante A, Mendoza-Flores R, Gosset G, Bolivar F. The aminoshikimic acid pathway in bacteria as source of precursors for the synthesis of antibacterial and antiviral compounds. J Ind Microbiol Biotechnol. 2021 Dec 23;48(9-10):kuab053. doi: 10.1093/jimb/kuab053. PMID 34374768
- [Background] PSA-Screening in Schweden: Deutlich geringere Prostatakarzinom-Mortalitat. Aktuelle Urol. 2023 Feb;54(1):10. doi: 10.1055/a-1925-4156. Epub 2023 Feb 14. No abstract available. German. PMID 36787767
- [Background] Baron-Mendoza I, Del Moral-Sanchez I, Martinez-Marcial M, Garcia O, Garzon-Cortes D, Gonzalez-Arenas A. Dendritic complexity in prefrontal cortex and hippocampus of the autistic-like mice C58/J. Neurosci Lett. 2019 Jun 11;703:149-155. doi: 10.1016/j.neulet.2019.03.018. Epub 2019 Mar 15. PMID 30885632
- [Background] Chen B, Wang Z, Chen Z, Qu X, Fang X, Wang X, Ke G. Comparison of Two Surgical Approaches to Supination-External Rotation-Type Ankle Fractures. J Healthc Eng. 2022 Apr 11;2022:7726726. doi: 10.1155/2022/7726726. eCollection 2022. PMID 35444779
- [Background] Zhang DDQ, Sussman J, Dossa F, Jivraj N, Ladha K, Brar S, Urbach D, Tricco AC, Wijeysundera DN, Clarke HA, Baxter NN. A Systematic Review of Behavioral Interventions to Decrease Opioid Prescribing After Surgery. Ann Surg. 2020 Feb;271(2):266-278. doi: 10.1097/SLA.0000000000003483. PMID 31356268